CLINICAL TRIAL: NCT03626246
Title: Pathogenesis of Compromised Bone Quality and Mechanics in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas Nickolas, MD MS, Associate Professor of Medicine, Columbia University
Other Study IDs: AAAQ7778; 1R01DK110871-01 (NIH)
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Chronic Kidney Disease; End Stage Kidney Disease; Chronic Kidney Disease Mineral and Bone Disorder; Renal Osteodystrophy; Secondary Hyperparathyroidism
Keywords: Bone loss; Bone fracture; Bone biopsy; Kidney
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder; Hyperparathyroidism, Secondary; Bone Diseases, Metabolic; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We would like to store the biological samples that you agreed to provide as part of this study: Blood, bone, urine and muscle.
  DNA taken from these samples and/or the data obtained from the study and possibly use them for future research. They will be stored at CUMC either with the researchers on this study or in a central storage facility called a repository.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney disease: Patients who participate in our study are 40 years old or older and have a Chronic kidney disease stage 3, 4 or 5.
  Interventions: Other: Kidney disease

INTERVENTIONS:
Other: Kidney disease — Being part of this study you agree to participate in all these interventions:
  Genetic:
  • Blood sample
  Procedure/Surgery:
  • Bone and muscle biopsies.
  Radiation:
  * Bone density (DXA)
  * Thoracic and lumbar spine plain films.
  * HRpQCT: high-resolution peripheral quantitative computed tomography
  Other:
  * Completing medical history, physical activity level, and dietary questionnaires for calcium and vitamin D.
  * Measure levels of Advanced Glycation End products (AGEs) in the skin.

SUMMARY:
Kidney disease patients have a variety of bone disorders that result in bone loss and fractures. The mechanisms of these bone disorders are not clear but may be related to abnormal modification of a bone protein known as collagen. Therefore, the investigators are conducting this research study to identify underlying mechanisms that are responsible for the disruption of bone collagen and determining whether the abnormal bone collagen impairs bone strength. The investigators intend to identify these mechanisms through studying relationships between kidney disease and bone strength via bone imaging, bone biopsy and non-invasive measures from blood and skin.

DETAILED DESCRIPTION:
Kidney disease patients have abnormal protein (bone collagen) modifications in their bone that may increase the risk of breaking a bone (fracture). Preventing bone collagen from becoming abnormal may decrease the risk of breaking a bone, such as the spine or hip. Currently, the effect of abnormal bone collagen on bone strength is not fully defined, and there are no methods to measure the abnormal protein content without a bone biopsy. The purpose of this study is to define the effects of bone collagen on bone strength and to identify non-invasive markers that will tell us how much abnormal collagen is in the bone. If the investigators are able to identify a non-invasive marker of abnormal bone protein then they may be able to prevent the build-up of this protein and lower the risk of a fracture.

If the participant chooses to be in the study, the investigators will get information from the participant's medical records such as diagnosis, the medicines and treatments prescribed by the participant's doctor, and the participant's lab test results.

There will be two study visits, each lasting about 3 hours.

Visit 1: At the baseline visit, study procedures include:

* Completing medical history, physical activity level, and dietary questionnaires for calcium and vitamin D.
* Blood sample
* Bone Imaging will: dual energy X-ray absorptiometry (DXA) to measure bone mineral density, high-resolution peripheral quantitative computed tomography (HRpQCT) to measure bone quality, and back x-rays to assess for the presence of spine fractures.Females who are able to become pregnant will also provide a urine specimen for pregnancy testing. (A negative pregnancy test is required prior to bone imaging.)
* Measure levels of Advanced Glycation End products (AGEs) in the skin of the participant's forearm and also in the participant's bone by bone biopsy. Advance Glycation End products may play a role in the development of weakened bone due to chronic kidney disease.

Visit 2: The participant's second visit will occur within 6-months of enrollment. At this visit, the participant will undergo a bone and muscle biopsy at the hip area under conscious sedation and a localized pain numbing medicine. The bone biopsy provides detailed information about the quality of the participant's bone that cannot be obtained through other tests like x-rays or blood tests. The investigators will use the bone biopsy to determine the amount of abnormal protein in the participant's bone. The muscle biopsy informs about the health of the participant's muscle fibers and allows us to detect any muscle mass wasting associated to chronic kidney disease. Since the piece of muscle is taken form the bone biopsy, no extra incision is needed.

The duration of the participant's participation from start of antibiotics through the actual bone biopsy will be approximately 3 weeks and 5 days (26 days).

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 3, 4 or 5
* Stable dose of vitamin D for 2-months

Exclusion Criteria:

* Dialysis
* Current use or treatment in the past one year with oral or inhaled glucocorticoids for more than 90 days.
* Current use or treatment in the past one year with sex hormone/SERM therapy for more than 30 days.
* Any use of bisphosphonates.
* Use of anti-osteoporosis therapies (denosumab, teriparatide, calcitonin or anti-sclerostin antibodies) in last 2 years.
* Any solid organ transplant or bone marrow transplant (Not including skin or cornea).
* Patients on non-aspirin anticoagulants that cannot be reasonably held for biopsy.
* Any cancers within 5-yrs of diagnosis that were metastatic to bone, and that are not in complete remission
* Any history of leukemia, multiple myeloma, lymphoma, amyloid or paraproteinemias.
* Any congenital or acquired collagen of bone diseases other than osteoporosis or renal osteodystrophy (Including but not limited to: Osteogenesis Imperfecta, X-Linked Hypophosphatemic Rickets, Pagets or Cushings Disease).
* History of Primary Hyperparathyroidism within 2-years of Parathyroidectomy.
* Hypoparathyroidism - primary or post-surgical
* Hyperthyroidism - if untreated and not on stable dose of medication for 6 months
* Hypothyroidism - if untreated and not on stable dose of medication for 6 months
* Non-ambulatory
* Bilateral lower extremity amputations.
* Weight >300 lbs.
* Medical disease - end stage heart, end stage liver, celiac disease and other intestinal malabsorption

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the general nephrology clinics at Columbia University Medical Center. Subjects referred for both clinical biopsy and those only participating in the research protocol will be eligible. The main clinical indication for bone biopsy in CKD patients is to determine turnover status for selection of type of bone active agent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Determine amounts of abnormal collagen present in the bone of CKD patients | 2.5 years
  In patients with CKD stage 3-5, the investigators will obtain transiliac crest bone biopsies and determine the amount of advanced glycation end-products that are present in bone collagen
Determine if greater amounts of abnormal collagen in the bone of CKD patients decreases bone strength | 1 year
  In patients with CKD stage 3-5, the investigators will perform biomechanical testing of bone biopsy specimens and determine if greater degree of advanced glycation end-product modification of bone collagen changes bone strength.
To identify non-invasive biomarkers of advanced glycation end-products in bone collagen | 1 year
  In patients with CKD stage 3-5, to obtain blood and skeletal imaging with high resolution peripheral computed tomography and to determine if the concentration of advanced glycation end-products in bone collagen can be identified by non-invasive methods.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nickolas, MD,MS, Principal Investigator — Columbia University
Locations (1):
- Columbia/CUMC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided